CLINICAL TRIAL: NCT04018443
Title: The Relation Between Common Carotid Artery Diameter and Central Venous Pressure for Assessment of Intravascular Fluid Status After Major Surgeries: An Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa A. Kasem, Associate professor, Beni-Suef University
Other Study IDs: FM-BSU REC: 007/2019
Record Dates: First submitted 2019-07-07; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Fluid Resuscitation Monitoring Non-invasively

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients admitted ti surgical ICU after major surgery: patient admitted to surgical ICU after major surgery for post-operative close monitoring, assessment and resuscitation of the intravascular volume status
  Interventions: Diagnostic Test: common carotid artery diameter measurement

INTERVENTIONS:
Diagnostic Test: common carotid artery diameter measurement — measurement of common carotid artery diameter will be carried out two times: the initial measurement (pre-infusion) which is followed by infusion of crystalloid solution (Ringer lactate) 30 ml/min till reaching a total infusion volume of 7 ml/kg body weight then another ultrasound measurement will be taken (prost-infusion). Between these sequential measurements, the patient position will not be changed. The percentage increase in CCA diameter will be calculated using the formula: [(dia-mpost/dia-mpre) × 100] - 100 [11].

SUMMARY:
Recently, bedside ultrasound has become an important tool for the simple and non-invasive hemodynamic assessment of critically ill patients. This applies not only to echocardiography but also to ultrasound of large extra-thoracic veins. The sonography can provide real time assessment of the vascular system and hemodynamic status at the bedside.

To our knowledge, there is one report about the association between sonographically assessed carotid artery diameter and intravascular volume, which raised recommendation for further studies including the interplay between carotid geometry and intravascular fluid status.

Aim of the study:

The aim of this work is to evaluate the accuracy of noninvasive techniques for assessment of intravascular volume status by Sonographic assessment of both the common carotid artery diameter (CCA) and the central venous pressure (CVP) in response to a bolus of crystalloid solution infusion and to find the correlation between CCA diameter and CVP as the primary outcome in adults patients after major surgeries who needs close assessment and maintenance of the intravascular volume status.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients (age 20-60 years).
2. ASA physical status I and II
3. Patients who are able to breathe spontaneously and lie supine.
4. Patients who have CVP catheter (subclavian or internal jugular vein).

Exclusion Criteria:

1. History of carotid artery surgery
2. Significant cardiac disease (cardiomyopathy and/or moderate to severe valvular heart lesion).
3. Significant hepatic disease (Child-Pugh score B or C ).
4. Renal failure.
5. Obesity: BMI ˃ 30 kg/m2
6. Need for mechanical ventilation.
7. Pregnancy.
8. Unstable vital signs during the process of sonography (e.g. the patients on vasoactive drugs)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients scheduled for elective or emergency major surgeries including, including (but not limited to) (abdominal exploration for intestinal obstruction or after trauma, aorto-femoral bypass, radical cystectomy, etc..) that require post-operative close monitoring, assessment and resuscitation of the intravascular volume status
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-07 (Actual); Primary Completion 2019-10-07 (Estimated); Study Completion 2019-10-07 (Estimated)

PRIMARY OUTCOMES:
Common Carotid Artery diameter at expiration (millimetre) | 30 minutes before fluid bolus infusion
  common carotid artery internal diameter changes songraphically measured to assess intravenous resuscitation
Common Carotid Artery diameter at expiration (millimetre) | 5 minutesafter fluid bolus infusion
  common carotid artery internal diameter changes songraphically measured to assess intravenous resuscitation
Central venous pressure (centimetre water) | 5 minutes after fluid bolus infusion
  Central venous pressure changes measured to assess intravenous resuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided